CLINICAL TRIAL: NCT06487260
Title: Mental Health and Symptoms of Energy Deficiency (REDs) in Young Biathletes.
Status: Completed | Type: Observational
Sponsor: Ostfold University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Inland Norway University of Applied Sciences (Other); International Biathlon Union (Unknown)
Responsible Party: Principal Investigator, Therese Fostervold Mathisen, Associate Professor, Ostfold University College
Other Study IDs: 733966
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue; Physical Health
Keywords: biathlon; biathletes; nordic skiing; REDs; LEA; Mental health; IBU; DXA; Eating Disorders; Blood work
MeSH Terms: conditions — Psychological Well-Being; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biathletes 16 years of age: Norwegian, competetive biathletes of both sexes, aged 16 years of age
- Biathletes 17 years of age: Norwegian, competetive biathletes of both sexes, aged 17 years of age
- Biathlete 18 years of age: Norwegian, competetive biathletes of both sexes, aged 18 years of age

SUMMARY:
Participation in weight-sensitive sports has been identified as a significant risk factor for low energy availability (LEA), relative energy deficiency in sport (REDs), and eating disorders. However, there is limited knowledge regarding the symptoms of LEA, REDs, and mental health issues in young biathletes. This study investigates the prevalence of these symptoms in young, talented biathletes from one of the leading nations in the sport. By including athletes of both sexes aged 16, 17, and 18, this study aim to determine whether symptom severity is associated with age, sex, or performance level. Furthermore, this study will explore the experiences of biathletes aged 18 and older with the new best practice guidelines for body composition assessment, designed by an IOC working group on the REDs consensus update of 2023 to safeguard athletes from negative experiences. The insights gained from this study may enhance the understanding of the frequency of health symptoms, the age or performance level at which symptoms typically increase, and the specific needs of athletes to ensure their safety and well-being in the sport.

DETAILED DESCRIPTION:
Being physically active is associated with a range of positive mental, physical, and psychosocial health benefits. Although athletes might be expected to enjoy these positive health effects, studies also show that high-level competitive athletes have a similar prevalence of certain mental disorders as the general population. Beyond reflecting the normal occurrence of mental health challenges in the population, performance expectations related to participation in competitive sports may contribute to many athletes experiencing periods or persistent mental health issues. Despite the increased openness in recent years about top athletes experiencing mental stress and disorders, there is little knowledge about the overall prevalence, especially among younger athletes at sub-elite performance levels. In 2023, Norwegian media highlighted a serious concern about the mental health of young biathletes, underscored by an alarming and unexpectedly high incidence of suicide among young biathlon talents.

Ski sports are among many weight-sensitive sports challenged by a high prevalence of eating disorders, particularly among female athletes. Eating disorders are linked to a high risk of low energy availability (LEA) and the syndrome relative energy deficiency (REDs) in athletes. REDs involve a variety of health challenges that follow LEA, and mental health issues can be both contributing factors to and effects of LEA. Knowledge about the prevalence of LEA, eating disorders, and REDs specifically among biathletes is very limited. A recent study found that a group of young female skiers (17 years old), including biathletes, on average consumed too little energy and carbohydrates relative to their athletic needs, and that 17% had LEA. A previous study recruited female athletes aged 25 years with self-expressed concern for REDs. This study found an overall prevalence of eating disorders corresponding to 21.3%, and that 65% in the sub-group of biathletes had LEA. Athletes with LEA symptoms had both lower weight and BMI, and the highest prevalence of eating disorders. At the same time, there is a study with young male skiers (including biathletes) aged 16 years, which finds a high prevalence of low bone mass and loss of bone mass through puberty. Low bone mass is one of the cardinal signs of LEA and REDs.

There is a need to map the prevalence of mental health issues and symptoms of REDs in young biathletes. Such knowledge can be used to understand the extent, specific vulnerable periods, and potentially explain why some are more affected than others. This knowledge can be used to more easily identify those who may need help and to initiate early interventions before the severity and complexity increase. In this exploratory national cross-sectional study, the aim is to map mental health and symptoms of REDs in young biathlon talents aged 16-19 years. In connection with mapping the physical symptoms of REDs, this study also aim to evaluate athlete experiences when closely following the new proposed guidelines and recommendations for measuring body composition in athletes. The guidelines (three members of this project group contributed in producing those guidelines) were given to protect athletes from negative experiences with body evaluation, so fewer are at risk of developing a negative body image and disordered eating behaviors or eating disorders.

This study works from the following hypotheses: 1) The prevalence of body dissatisfaction, depression, eating disorders, and symptoms of REDs (hereafter: outcome measures) is low in 16-year-old biathletes; 2) the prevalence of outcome measures increases with age and is therefore higher in 18-year-old biathletes; 3) the prevalence of eating disorders and symptoms of REDs is higher in girls than boys in all age groups; 4) young biathletes aged 18 years experience a professional and safe implementation of body composition evaluation when recommended guidelines are followed.

ELIGIBILITY:
Inclusion Criteria:

* competetive biathlete
* live in Norway, speaks or understand written and oral Norwegian

Exclusion Criteria:

* injured and prevented from regular training (3 months leading up to recruitement)

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young, competetive biathletes in age-range 16-20 years of age, living in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Eating Disorder | September 2024
  Number of athletes with a diagnosable eating disorder, and type of eating disorder. Evaulation will be by a clinical interview following the validated Eating Disorder Examination Inverview.
Symptom of Eating Disorders | September 2024
  Number of athletes with symptoms of eating disorders, and type of eating disorder. Evaulation will be by a selfreport responding to the Eating Disorder Examination Questionnaire.
Symptoms of Depression | September 2024
  Severity in symptoms of depression and number of athletes with symptoms of depression. Evaulation will be by selfreport, responding to the Beck Depression Inventory v-2
Symptoms of Low Energy Availability (LEA) | September 2024
  Severity in symptoms of LEA, evaluated by selfreport, responding to the Low Energy Availability for Females Questionnaire, and Low Energy Availiability for males Questionnaire.
Body composition | September 2024
  Body composition (fat mass and lean body mass) measured by DXA, as part of the evaluation of fitness in biathletes 18 years or older
Bone mineral Density | September 2024
  Bone mineral density in biathletes 18 years or older, as a fitness evaluation and symptom of LEA

SECONDARY OUTCOMES:
Blood work, energy metabolism | September 2024
  Hormone T3 measured by blood sample to evaluate energy metabolism as a symptom of LEA
Blood pressure, orthostatic | September 2024
  The orthostatic blood pressure, as a symptom of LEA
Blood pressure, resting | September 2024
  The resting blood pressure, as a symptom of LEA
Resting heart rate | September 2024
  Resting heart rate, as a measure of cardiovascular fitness and symptom of LEA
Indirect calorimetry | September 2024
  Indirect calorimetry as a measure of energy metabolism, serving as a symptom of energy availability

OTHER OUTCOMES:
Body appreciation | September 2024
  Evaulation of body appreciation by the Body Appreciation Scale (BAS, version 2), as a measure for protective/posiitive trait versus risk for Eating Disorders
Blood work, iron status | September 2024
  Serum ferritin, transferrin, and serum-iron will be measured as a complete evaluation of iron status
Blood work, cholesterol | September 2024
  Total cholesterol and low density lipoprotein (LDL cholesterol) will be measured for evaulation of health and symptoms of LEA
Experience from body composition assessment | September 2024
  Interview of biathletes 18 years or older who participate in DXA measurements. Focus is on how they experience the total body composition assessment as we follow the best practice guidlines. Interview is based on a semi-structured interview guide.
Demographics | September 2024
  Demographic description of the biathletes (age, competition level, training volume, history of bone fractures, history of menstrual cycle, history of any eating disorder diagnosis)
Urinary incontinence | September 2024
  Question on experience with urinary incontinence, as a symptom of LEA. Question is a yes/no response to any experience, and a positive response is further detailed about context (urge or stress)

CONTACTS AND LOCATIONS:
Overall Officials: Therese F Mathisen, PhD, Principal Investigator — Associate Professor
Locations (2):
- Norway (2):
  - Inland Norway University of Applied Sciences, Lillehammer, Inland
  - Norwegian School of Sport Sciences, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Undisclosed data can be shared upon reasonable request.
Time Frame: Available after 31.12.2025
Access Criteria: Any researcher that contacts the project group with a reasonable request (e.g. need of data for review, metaanalyses etc)